CLINICAL TRIAL: NCT06057649
Title: Effects of Effleurage Abdominal Massage on Pain and Quality of Life in Primary Dysmenorrhea Among Female University Students in Lahore
Brief Title: Effects of Effleurage Abdominal Massage on Pain and Quality of Life in Primary Dysmenorrhea Among Students in Lahore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Aqeela Sarwar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ION UHS
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; Female university students; Pain; Quality of Life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to control and experimental group. participants in control group will continue with their routine care and experimental group will receive effleurage abdominal massage alongwith routine practices
Who Masked: Outcomes Assessor
Masking Description: a third person will be involved as second assessor for blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): participants of control group will receive no intervention. they will be instructed to continue with their routine practices
- experimental (Experimental): Participants of experimental group will perform effleurage abdominal massage
  Interventions: Other: Effleurage Abdominal Massage

INTERVENTIONS:
Other: Effleurage Abdominal Massage — perform the effleurage massage by following these steps: Lie in supine position with knee slightly flexed. Start from the right lower quadrant, using gentle pressure, rub in tiny clockwise circular motions using any non-analgesic cream, towards right rib cage then towards upper left side, moving down the left side to hip bone. Keep up the circular massage while moving inward, toward your belly button for three minutes. After three minutes, use a little more pressure, continuing the circular movements for 10 minutes. Massage for 10 minutes a day for two months during the first 3 days of the menstrual cycle.
  Arms: experimental

SUMMARY:
To find out the answer of the study question that effleurage abdominal massage has any effect on pain and quality of life in primary dysmenorrhea among university students or nota study will be conducted with an objective to evaluate the effects of effleurage abdominal massage on pain and quality of life in primary dysmenorrhea among university students

DETAILED DESCRIPTION:
Primary dysmenorrhea, the commonly occurring gynecological issue faced by young girls. It severely affects quality of female life. It leads to fatigue, psychological issues, lack of interest in selfcare and daily activities that results in absenteeism at work and educational institutes. It also badly affects academic performance and extra-curricular activities. Different pharmacological and non-pharmacological interventions are being used for reducing its negative effects, such as effleurage abdominal massage intend to decrease the problems faced by students as a result of this frightening issue. Here the question arises for health professionals that effleurage abdominal massage has any effect on pain and quality of life in primary dysmenorrhea among university students or not? To find out the answer of this question a study will be conducted with an objective to evaluate the effects of effleurage abdominal massage on pain and quality of life in primary dysmenorrhea among university students. This study holds considerable implications in addressing potential adverse effects associated with pharmacological analgesic agents, thereby mitigating pain, lack of interest in work and enhancing functional capacity, hence improving quality of life. Moreover, it is anticipated to contribute to the reduction of healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried female university students from Lahore
* Aged between 18-25 years
* Diagnosed patients by gynecologist with primary dysmenorrhea for three previous consecutive cycles.
* Regular menstrual cycles ranging 21-35 days lasting for 3-7 days.
* Having pain score of 6 or more than 6 on Numeric Pain Rating Scale

Exclusion Criteria:

* Presence of any known abdominal or pelvic disease.
* Obstructive vaginal or uterine congenital anomalies.
* Presence of known or suspected secondary dysmenorrhea.
* History of major abdominal or pelvic surgery in the previous three months.
* History of hormonal therapy in the last six months.
* History of using analgesics during menstruation.
* History of having any medical disease i.e. cardiac and renal disease.
* Participants doing regular exercise.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primary dysmenorrhea belongs to female gender
Enrollment: 52 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Dysmenorrhea Induced Pain intensity | 3 months
  Outcome Measurement Tool:
  Numeric Pain Rating Scale:
  Dysmenorrhea induced pain intensity measured by Numerical pain rating scale will be used having numbers from 0 to 10 to indicate the intensity of pain. Here is a breakdown of the numeric rating pain scale
  * 0: No pain.
  * 1-3: Mild pain.
  * 4-6: Moderate pain.
  * 7-9: Severe pain.
  * 10: Excruciating pain.
Measure the level of Quality of Life | 3 months
  Outcome Measurement Tool:
  Euroqol-5D-5L scale for Quality of Life:
  The EQ-5D-5L scale will be used to assess students' quality of life across five dimensions and will allow respondents to indicate their level of functioning or health in each dimension with 1 as highest and 5 as lowest for each dimension. Additionally, EQ-5D-5L includes a visual analog scale (VAS) that will allow respondents to rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Aqeela Sarwar, MS Nursing, Study Chair — PG Nursing
Locations (1):
- College of Nursing AIMC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No